CLINICAL TRIAL: NCT02128100
Title: The Effect of FOLFIRINOX and Stereotactic Body Radiation Therapy for Locally Advanced, Non-Resectable Pancreatic Cancer
Brief Title: Effects of Folfirinox and Stereotactic Body Radiation Therapy for Advanced Pancreatic Cancer
Acronym: BCC-RAD-13
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Neal Edward Dunlap, Associate Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14.0413
Record Dates: First submitted 2014-04-22; First posted 2014-05-01 (Estimated); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Pancreatic Cancer Non-resectable
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Folririnox with SBRT (Experimental): Folfirinox
  * Oxaliplatin 85 mg/m² for over 2 hours,
  * Leucovorin 400n mg/m² for over 2 hours,
  * Irinotecan 180 mg/m² for over 90 minutes, along with Leucovorin infusion
  * Fluorouracil 400 mg/m² as a fast infusion over 15 minutes
  * Fluorouracil 2400 mg/m² as a slow infusion over 46 hours
  SBRT 5 treatments of stereotactic body radiation therapy (SBRT) over the course of two weeks with a minimum of 36 hours in between each treatment.
  Interventions: Drug: Folfirinox; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Folfirinox — * Oxaliplatin 85 mg/m² for over 2 hours,
  * Leucovorin 400n mg/m² for over 2 hours,
  * Irinotecan 180 mg/m² for over 90 minutes, along with Leucovorin infusion
  * Fluorouracil 400 mg/m² as a fast infusion over 15 minutes
  * Fluorouracil 2400 mg/m² as a slow infusion over 46 hours
  Other Names: o Oxaliplatin; o Leucovorin; o Irinotecan; o Fluorouracil
Radiation: Stereotactic Body Radiation Therapy — 5 treatments of stereotactic ablative radiotherapy (SABR) over the course of two weeks with a minimum of 36 hours in between each treatment.

SUMMARY:
This study wants to find out how safe and effective the use of Folfirinox combined with Stereotactic Body Radiation Therapy )(SBRT) is for the treatment of pancreatic cancer.

DETAILED DESCRIPTION:
The study will be a prospective, non-randomized, single center, trial to assess the effects of FOLIRINOX chemotherapy with SBRT on locally advanced, non-resectable pancreatic cancer. Patients will either undergo a biopsy to confirm the diagnosis or have strong clinical suspicion of a new cancer or recurrence based on the recommendations of a multi-disciplinary GI oncology team. FOLFIRINOX with be delivered prior to SBRT for 4 cycles. Restaging imaging will occur prior to SBRT delivery. SBRT will be delivered using standard stereotactic techniques to a dose of 3200cGy at 650cGy per fraction delivered over 2 weeks. Additional adjuvant chemotherapy with be delivered at the physician's discretion. Patients will be reassessed both clinically and radiographically at 3 months, 6 months, 9 months and 12 months post-treatment. Quality of life analysis will occur at 3 month intervals after treatment. Blood will be drawn for exploratory biomarker analysis at strategic timepoints during treatment and followup. Following the initial imaging time points, standard surveillance will be employed with clinical assessment and imaging at 3 month intervals for the first 2 years post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* ECOG performance status 0-1
* Pathologic or clinical diagnosis of a new pancreatic adenocarcinoma. A reasonable attempt should be made to make a pathologic diagnosis of malignancy.
* Imaging as follows:

  * CT scan of the chest, abdomen and pelvis with IV and oral contrast within 8 weeks of registration
  * Whole body PET scan within 8 weeks of registration
* Evaluation by a surgical oncologist to determine non-resectability
* Negative serum pregnancy test within 2 weeks prior to registration for women of childbearing potential.
* CBC/differential obtained within 14 days prior to registration with adequate bone marrow function as follows:

  * ANC > 1,500 cell/mm3
  * Platelets > 100,000 cells/mm3
  * Hemoglobin > 8.0 g/dl (transfusion to obtain this value is permissible)
* Additional labs within 14 days prior to registration

  * CA 19-9
  * Creatinine <2mg/dl
  * Bilirubin <2mg/dl
  * AST and ALT < 2.5 x ULN
* Patients must provide study specific informed consent prior to study entry.

Exclusion Criteria:

* Metastatic disease as defined by the multi-disciplinary team
* Prior anti-cancer therapy for a pancreatic tumor
* Prior malignancy within the last 3 years.
* Pregnant women or lactating women
* Acquired Immune Deficiency Syndrome (AIDS) based on CDC criteria. However HIV testing is not manditory for this protocol
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-09-19 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal E Dunlap, MD, Principal Investigator — James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Folririnox With SBRT: Folfirinox Oxaliplatin 85 mg/m² for over 2 hours, Leucovorin 400n mg/m² for over 2 hours, Irinotecan 180 mg/m² for over 90 minutes, along with Leucovorin infusion Fluorouracil 400 mg/m² as a fast infusion over 15 minutes Fluorouracil 2400 mg/m² as a slow infusion over 46 hours
  SBRT 5 treatments of stereotactic body radiation therapy (SBRT) over the course of two weeks with a minimum of 36 hours in between each treatment.
  Folfirinox:
  Oxaliplatin 85 mg/m² for over 2 hours, Leucovorin 400n mg/m² for over 2 hours, Irinotecan 180 mg/m² for over 90 minutes, along with Leucovorin infusion Fluorouracil 400 mg/m² as a fast infusion over 15 minutes Fluorouracil 2400 mg/m² as a slow infusion over 46 hours
  Stereotactic Body Radiation Therapy: 5 treatments of stereotactic ablative radiotherapy (SABR) over the course of two weeks with a minimum of 36 hours in between each treatment.
Period: Overall Study
Arm/Group | Folririnox With SBRT
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Folririnox With SBRT: Folfirinox
  * Oxaliplatin 85 mg/m² for over 2 hours,
  * Leucovorin 400n mg/m² for over 2 hours,
  * Irinotecan 180 mg/m² for over 90 minutes, along with Leucovorin infusion
  * Fluorouracil 400 mg/m² as a fast infusion over 15 minutes
  * Fluorouracil 2400 mg/m² as a slow infusion over 46 hours
  SBRT 5 treatments of stereotactic body radiation therapy (SBRT) over the course of two weeks with a minimum of 36 hours in between each treatment.
  Folfirinox: o Oxaliplatin 85 mg/m² for over 2 hours,
  * Leucovorin 400n mg/m² for over 2 hours,
  * Irinotecan 180 mg/m² for over 90 minutes, along with Leucovorin infusion
  * Fluorouracil 400 mg/m² as a fast infusion over 15 minutes
  * Fluorouracil 2400 mg/m² as a slow infusion over 46 hours
  Stereotactic Body Radiation Therapy: 5 treatments of stereotactic ablative radiotherapy (SABR) over the course of two weeks with a minimum of 36 hours in between each treatment.
Arm/Group | Folririnox With SBRT
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Grade 3 or Higher Adverse Event(s) as a Measure of Safety and Tolerability
Description: Number of Participants With Grade 3 or Higher Adverse Event(s) as a Measure of Safety and Tolerability. This is based on CTCAE to assess toxicity at specified time points by the treating physician.
Time Frame: Assessed up to 24 months post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Folririnox With SBRT
Number analyzed (Participants) | 5
Participants | 3

2. Secondary Outcome: Overall Response Rate for Participants as Assessed by Contrast-enhanced CT Scan of the Abdomen at 12 Months.
Description: Response to therapy at 12 months post treatment as measured from CT Scan by modified RECIST criteria as follows; Response is measured as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum of LD.
Time Frame: Assessed at 3 months, 6 months, 9 months and 12 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Folririnox With SBRT
Number analyzed (Participants) | 4
Participants | 2

3. Other Pre Specified Outcome: Quality of Life Assessment at 12 Months Post-treatment
Description: Assessment is based on participant results from administration of the Functional Assessment of Cancer Therapy - Pancreas (FACT-Hep). FACT-Hep is an established tool for measuring quality of life both before and after intervention. The form consists of 45 questions and should take approximately 8 minutes to complete. Higher scores indicate higher quality of life. This assessment consists of the following sub-scales (with associated score ranges): Physical Well-Being (0-28); Social/Family Well-Being (0-28); Emotional Well-Being (0-24); Functional Well-Being (0-28); Hepatobiliary Cancer (0-72). All items are ranked on a five-point scale ranging from 0-4. Results were based on the mean FACT-G total score of all participants. The FACT-G total score is derived from the sum of scores on the Physical, Emotional, Social/Family, Functional Well-Being and Hepatobiliary Cancer subscales and is designed to measure Health Related Quality of Life (HRQOL) in subjects undergoing cancer treatment.
Time Frame: 12 months from completion of therapy
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Folririnox With SBRT
Number analyzed (Participants) | 4
score on a scale | 115 (12)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Folririnox With SBRT
All-Cause Mortality (participants affected / at risk) | 3/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Folririnox With SBRT (N=5)
Hypokalemia (Metabolism and nutrition disorders) | 1 — CTCAE grade 1 = 1
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 3 — CTCAE grade 1 = 2 patients, grade 2 = 1 patient (all resolved)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-09-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT02128100/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT02128100/ICF_001.pdf